CLINICAL TRIAL: NCT03988842
Title: Standard-dose Apixaban AFtEr Very Low-dose ThromboLYSis for Acute Intermediate-high Risk Acute Pulmonary Embolism
Acronym: SAFE-LYSE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Victor Tapson, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Victor Tapson, MD, Director, Clinical Research for the Women's Guild Lung Institute; Director, Venous Thromboembolism and Pulmonary Vascular Disease Research Program; Associate Director, Pulmonary and Critical Care Division, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00054951
Record Dates: First submitted 2019-05-24; First posted 2019-06-18 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Embolism With Acute Cor Pulmonale; Pulmonary Embolism; Pulmonary Embolism With Pulmonary Infarction; Pulmonary Embolism Subacute Massive; Right Ventricular Dysfunction; Right Ventricular Failure
MeSH Terms: conditions — Pulmonary Embolism; Ventricular Dysfunction, Right; Heart Failure | interventions — Tissue Plasminogen Activator; Heparin; apixaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alteplase & Unfractionated Heparin & Apixaban (Experimental): Alteplase 24mg intravenous infusion for 20 minutes followed by unfractionated heparin intravenous infusion over 24 hours followed by apixaban 10mg tablet twice-daily for one week followed by apixaban 5mg tablet twice-daily for at least 6 months.
  Interventions: Drug: Alteplase; Drug: Unfractionated heparin; Drug: Apixaban
- Placebo & Unfractionated Heparin & Apixaban (Active Comparator): Alteplase placebo solution 24mg intravenous infusion for 20 minutes followed by unfractionated heparin intravenous infusion over 24 hours followed by apixaban 10mg tablet twice-daily for one week followed by apixaban 5mg tablet twice-daily for at least 6 months.
  Interventions: Drug: Unfractionated heparin; Drug: Placebo; Drug: Apixaban

INTERVENTIONS:
Drug: Alteplase — Lyophilized powder for reconstitution in 50mg vials
  Other Names: Activase; tissue-type plasminogen activator
  Arms: Alteplase & Unfractionated Heparin & Apixaban
Drug: Unfractionated heparin — Heparin sodium in 0.45% sodium chloride injection for intravenous use
  Other Names: Heparin sodium
Drug: Placebo — Saline solution reconstituted to mimic Alteplase 50mg vial
  Other Names: Placebo (for Alteplase)
  Arms: Placebo & Unfractionated Heparin & Apixaban
Drug: Apixaban — Apixaban tablet
  Other Names: Eliquis

SUMMARY:
The purpose of this study is to examine the degree to which pulmonary embolism (clot) can be dissolved when treated with a very low dose of a systemic thrombolytic drug (clot buster) along with standard anticoagulant therapy as compared to the standard of care anticoagulant therapy alone.

DETAILED DESCRIPTION:
The OVERALL OBJECTIVE of this investigation is to determine whether very low-dose intravenous tissue-type plasminogen activator [tPA] (24 mg) + standard anticoagulation therapy (intravenous heparin) for treatment of acute PE (pulmonary embolism) in intermediate-high risk patients will have superior clot lysis (breakdown of clot) by chest CTA (computed tomography angiography) at 24 ± 6 hours post infusion compared to standard of care treatment alone. Acute intermediate-high risk PE patients are those with acute symptoms <14 days), simplified Pulmonary Embolism Severity Index (sPESI)>0, normal systemic arterial blood pressure (>90mmHg) without vasopressor support, elevated biomarkers (troponin or BNP), and evidence of RV dysfunction (right ventricular to left ventricular ratio>0.9).The study is planned to evaluate the reduction in clot burden based on the obstruction index using the Refined Modified Miller Score (RMMS), improvement in right ventricular (RV) function, and overall safety in the two treatment groups. 40 Subjects with intermediate-high risk PE (hemodynamically stable PE with a RV/LV ratio ≥ 0.9, elevated biomarkers, and sPESI>0) will be recruited and randomized to one of two treatment groups: 24mg of systemic (IV) tPA + IV unfractionated heparin versus saline placebo + IV unfractionated heparin. After delivery of the systemic (IV) tPA/placebo, patients will continue IV unfractionated heparin therapy for at least 24 hours. If there is no evidence of active bleeding nor significant hemoglobin drop (i.e., ≥ 2 mg/dL), patients will be transitioned to standard dose apixaban, 10 mg twice-daily x one week followed by 5 mg twice-daily for at least 6 months. Some patients will require indefinite apixaban therapy based on patient-specific factors, including unprovoked nature of PE event, and/or persisting DVT/PE risk factors. Finally, consideration will be given for decreasing the apixaban dose to 2.5 mg twice-daily after 6 months. Apixaban was selected as the anticoagulant of choice due to its very favorable bleeding profile in large clinical trials, which is an important consideration when prescribing an anticoagulant following systemic thrombolysis. Within 24 ± 6 hours post study drug infusion, a repeat chest CTA and echocardiogram will be performed. sPESI will also be calculated at this timepoint.At Day 30, 180 and 365, all subjects will have clinic visits which will include a physical exam, repeat echocardiogram if previous echo was abnormal, 6 minute walk test (6MWT), quality of life questionnaires, assessment of adverse and bleeding events and a review of concomitant medications including compliance with apixaban. At Days 3, 7, 90 and 270, a remote health check will occur via telephone or email assessing adverse and bleeding events, alongside a review of concomitant medications (including an assessment of compliance with apixaban).The standard of care for patients with submassive PE is to either receive anticoagulant therapy, EKOS (Catheter Assisted Thrombolysis) or thromboectomy. tPA is given at the FDA approved dose (100mg) occasionally at doses much higher than our study proposes. PatientS with PE will have the initial CTA, echocardiogram and lab work as standard of care. The follow up CTA is usually standard of care at Day 30 and the follow up echocardiograms are considered standard of care if the previous echocardiogram was abnormal.The study is being done as a proof of concept that low dose tPA is effective in clot lysis and will result in far less risk than the FDA dose. If our study achieves its aims, the research will advance clinical practices in treating pulmonary embolism by reporting the safety of lower dose tPA and opening opportunities to further explore the use of lower dose tPA to improve patient safety and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Chest CT angiogram (CTA) evidence of proximal Pulmonary Embolism (PE) with a filling defect in at least one main pulmonary artery or lobar artery
* PE symptom duration ≤14 days
* Intermediate-high risk PE: defined as RV dysfunction with an RV/LV diameter ≥ 0.9, sPESI > 0, and either troponin > 0.05ng/mL or BNP > 100 pg/mL, and hemodynamically stable (systolic blood pressure > 90mmHg without the use of vasopressor support)
* Randomization within 24 + 4 hours of anticoagulation
* Signed and dated informed consent obtained from subject or legally authorized representative before initiation of any study procedures

Exclusion Criteria:

* Weight > 130kg or < 40 kg on day of randomization
* Stroke or transient ischemic attack (TIA), head trauma, or other active intracranial or intraspinal disease within one year
* Recent (within one month) or active bleeding from a major organ
* Major surgery within 14 days
* Clinician deems the subject too high-risk for bleeding using HAS-BLED criteria
* History of any hematologic disease or coagulopathy
* Cirrhosis (as determined by Child-Pugh B or C)
* History of heparin-induced thrombocytopenia (HIT)
* Hemodynamic instability defined as systolic blood pressure (SBP) less than 90mmHg and/or use of vasopressors for greater than 15 minutes
* Severe hypertension as defined as SBP greater than 180mmHg
* Cardiac arrest or active cardiopulmonary resuscitation (CPR)
* Receiving neuraxial anesthesia or undergoing spinal puncture
* Patient with prosthetic heart valves
* Evidence of irreversible neurological compromise
* Evidence of poor functional status
* History of major gastrointestinal bleed within the last month
* Active gastric or duodenal ulcers
* Use of thrombolytics or glycoprotein IIb/IIIa antagonists within 3 days prior to diagnosis
* Lovenox administration within 12 hours of randomization
* Direct-acting oral anticoagulant use (dabigatran, rivaroxaban, apixaban, or edoxaban) with last known dose within 48 hours
* Hemoglobin < 10 g/dL
* Creatinine clearances < 60 mL/min
* Platelets < 100 thousand/µL
* INR > 1.4
* Alanine transaminase (ALT) or aspartate transaminase (AST) ≥ 2 times upper limit of normal (ULN)
* Total bilirubin (TBL) ≥ 1.5 times ULN (except due to confirmed Gilbert's syndrome)
* Patient is pregnant (positive pregnancy test; women of childbearing capacity must be tested prior to enrollment) or breast feeding
* Patient who is a prisoner, or if subject who becomes compulsory detained
* Active cancer defined as diagnosis of cancer within six months before the study inclusion, or receiving treatment for cancer at the time of inclusion or any treatment for cancer during 6 months prior to randomization, or recurrent locally advanced or metastatic cancer
* Known allergy, hypersensitivity or thrombocytopenia from heparin, tPA, or apixaban or iodinated contrast except for mild-moderate contrast allergies for which steroid pre-medication can be administered within 12 hours prior to the CTA
* HIV/AIDS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor F Tapson, MD, Principal Investigator — Cedars-Sinai Medical Center; Aaron S Weinberg, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Beckman MG, Hooper WC, Critchley SE, Ortel TL. Venous thromboembolism: a public health concern. Am J Prev Med. 2010 Apr;38(4 Suppl):S495-501. doi: 10.1016/j.amepre.2009.12.017. PMID 20331949
- [Background] Layish DT, Tapson VF. Pharmacologic hemodynamic support in massive pulmonary embolism. Chest. 1997 Jan;111(1):218-24. doi: 10.1378/chest.111.1.218. No abstract available. PMID 8996020
- [Background] Goldhaber SZ, Visani L, De Rosa M. Acute pulmonary embolism: clinical outcomes in the International Cooperative Pulmonary Embolism Registry (ICOPER). Lancet. 1999 Apr 24;353(9162):1386-9. doi: 10.1016/s0140-6736(98)07534-5. PMID 10227218
- [Background] Konstantinides SV, Torbicki A, Agnelli G, Danchin N, Fitzmaurice D, Galie N, Gibbs JS, Huisman MV, Humbert M, Kucher N, Lang I, Lankeit M, Lekakis J, Maack C, Mayer E, Meneveau N, Perrier A, Pruszczyk P, Rasmussen LH, Schindler TH, Svitil P, Vonk Noordegraaf A, Zamorano JL, Zompatori M; Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). 2014 ESC guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Nov 14;35(43):3033-69, 3069a-3069k. doi: 10.1093/eurheartj/ehu283. Epub 2014 Aug 29. No abstract available. PMID 25173341
- [Background] Kohn CG, Mearns ES, Parker MW, Hernandez AV, Coleman CI. Prognostic accuracy of clinical prediction rules for early post-pulmonary embolism all-cause mortality: a bivariate meta-analysis. Chest. 2015 Apr;147(4):1043-1062. doi: 10.1378/chest.14-1888. PMID 25317677
- [Background] Dalla-Volta S, Palla A, Santolicandro A, Giuntini C, Pengo V, Visioli O, Zonzin P, Zanuttini D, Barbaresi F, Agnelli G, et al. PAIMS 2: alteplase combined with heparin versus heparin in the treatment of acute pulmonary embolism. Plasminogen activator Italian multicenter study 2. J Am Coll Cardiol. 1992 Sep;20(3):520-6. doi: 10.1016/0735-1097(92)90002-5. PMID 1512328
- [Background] Meyer G, Vicaut E, Danays T, Agnelli G, Becattini C, Beyer-Westendorf J, Bluhmki E, Bouvaist H, Brenner B, Couturaud F, Dellas C, Empen K, Franca A, Galie N, Geibel A, Goldhaber SZ, Jimenez D, Kozak M, Kupatt C, Kucher N, Lang IM, Lankeit M, Meneveau N, Pacouret G, Palazzini M, Petris A, Pruszczyk P, Rugolotto M, Salvi A, Schellong S, Sebbane M, Sobkowicz B, Stefanovic BS, Thiele H, Torbicki A, Verschuren F, Konstantinides SV; PEITHO Investigators. Fibrinolysis for patients with intermediate-risk pulmonary embolism. N Engl J Med. 2014 Apr 10;370(15):1402-11. doi: 10.1056/NEJMoa1302097. PMID 24716681
- [Background] Chatterjee S, Chakraborty A, Weinberg I, Kadakia M, Wilensky RL, Sardar P, Kumbhani DJ, Mukherjee D, Jaff MR, Giri J. Thrombolysis for pulmonary embolism and risk of all-cause mortality, major bleeding, and intracranial hemorrhage: a meta-analysis. JAMA. 2014 Jun 18;311(23):2414-21. doi: 10.1001/jama.2014.5990. PMID 24938564
- [Background] Marti C, John G, Konstantinides S, Combescure C, Sanchez O, Lankeit M, Meyer G, Perrier A. Systemic thrombolytic therapy for acute pulmonary embolism: a systematic review and meta-analysis. Eur Heart J. 2015 Mar 7;36(10):605-14. doi: 10.1093/eurheartj/ehu218. Epub 2014 Jun 10. PMID 24917641
- [Background] Daley MJ, Murthy MS, Peterson EJ. Bleeding risk with systemic thrombolytic therapy for pulmonary embolism: scope of the problem. Ther Adv Drug Saf. 2015 Apr;6(2):57-66. doi: 10.1177/2042098615572333. PMID 25922654
- [Background] Kearon C, Akl EA, Ornelas J, Blaivas A, Jimenez D, Bounameaux H, Huisman M, King CS, Morris TA, Sood N, Stevens SM, Vintch JRE, Wells P, Woller SC, Moores L. Antithrombotic Therapy for VTE Disease: CHEST Guideline and Expert Panel Report. Chest. 2016 Feb;149(2):315-352. doi: 10.1016/j.chest.2015.11.026. Epub 2016 Jan 7. PMID 26867832
- [Background] Sors H, Pacouret G, Azarian R, Meyer G, Charbonnier B, Simonneau G. Hemodynamic effects of bolus vs 2-h infusion of alteplase in acute massive pulmonary embolism. A randomized controlled multicenter trial. Chest. 1994 Sep;106(3):712-7. doi: 10.1378/chest.106.3.712. PMID 8082346
- [Background] Goldhaber SZ, Agnelli G, Levine MN. Reduced dose bolus alteplase vs conventional alteplase infusion for pulmonary embolism thrombolysis. An international multicenter randomized trial. The Bolus Alteplase Pulmonary Embolism Group. Chest. 1994 Sep;106(3):718-24. doi: 10.1378/chest.106.3.718. PMID 8082347
- [Background] Wang C, Zhai Z, Yang Y, Wu Q, Cheng Z, Liang L, Dai H, Huang K, Lu W, Zhang Z, Cheng X, Shen YH; China Venous Thromboembolism (VTE) Study Group. Efficacy and safety of low dose recombinant tissue-type plasminogen activator for the treatment of acute pulmonary thromboembolism: a randomized, multicenter, controlled trial. Chest. 2010 Feb;137(2):254-62. doi: 10.1378/chest.09-0765. Epub 2009 Sep 9. PMID 19741062
- [Background] Zhang Z, Zhai ZG, Liang LR, Liu FF, Yang YH, Wang C. Lower dosage of recombinant tissue-type plasminogen activator (rt-PA) in the treatment of acute pulmonary embolism: a systematic review and meta-analysis. Thromb Res. 2014 Mar;133(3):357-63. doi: 10.1016/j.thromres.2013.12.026. Epub 2013 Dec 23. PMID 24412030
- [Background] Anderson CS, Robinson T, Lindley RI, Arima H, Lavados PM, Lee TH, Broderick JP, Chen X, Chen G, Sharma VK, Kim JS, Thang NH, Cao Y, Parsons MW, Levi C, Huang Y, Olavarria VV, Demchuk AM, Bath PM, Donnan GA, Martins S, Pontes-Neto OM, Silva F, Ricci S, Roffe C, Pandian J, Billot L, Woodward M, Li Q, Wang X, Wang J, Chalmers J; ENCHANTED Investigators and Coordinators. Low-Dose versus Standard-Dose Intravenous Alteplase in Acute Ischemic Stroke. N Engl J Med. 2016 Jun 16;374(24):2313-23. doi: 10.1056/NEJMoa1515510. Epub 2016 May 10. PMID 27161018
- [Background] Levine M, Hirsh J, Weitz J, Cruickshank M, Neemeh J, Turpie AG, Gent M. A randomized trial of a single bolus dosage regimen of recombinant tissue plasminogen activator in patients with acute pulmonary embolism. Chest. 1990 Dec;98(6):1473-9. doi: 10.1378/chest.98.6.1473. PMID 2123152
- [Background] Ucar EY. Update on Thrombolytic Therapy in Acute Pulmonary Thromboembolism. Eurasian J Med. 2019 Jun;51(2):186-190. doi: 10.5152/eurasianjmed.2019.19291. PMID 31258361
- [Background] Kucher N, Boekstegers P, Muller OJ, Kupatt C, Beyer-Westendorf J, Heitzer T, Tebbe U, Horstkotte J, Muller R, Blessing E, Greif M, Lange P, Hoffmann RT, Werth S, Barmeyer A, Hartel D, Grunwald H, Empen K, Baumgartner I. Randomized, controlled trial of ultrasound-assisted catheter-directed thrombolysis for acute intermediate-risk pulmonary embolism. Circulation. 2014 Jan 28;129(4):479-86. doi: 10.1161/CIRCULATIONAHA.113.005544. Epub 2013 Nov 13. PMID 24226805
- [Background] Piazza G, Hohlfelder B, Jaff MR, Ouriel K, Engelhardt TC, Sterling KM, Jones NJ, Gurley JC, Bhatheja R, Kennedy RJ, Goswami N, Natarajan K, Rundback J, Sadiq IR, Liu SK, Bhalla N, Raja ML, Weinstock BS, Cynamon J, Elmasri FF, Garcia MJ, Kumar M, Ayerdi J, Soukas P, Kuo W, Liu PY, Goldhaber SZ; SEATTLE II Investigators. A Prospective, Single-Arm, Multicenter Trial of Ultrasound-Facilitated, Catheter-Directed, Low-Dose Fibrinolysis for Acute Massive and Submassive Pulmonary Embolism: The SEATTLE II Study. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1382-1392. doi: 10.1016/j.jcin.2015.04.020. PMID 26315743
- [Background] Tapson VF, Sterling K, Jones N, Elder M, Tripathy U, Brower J, Maholic RL, Ross CB, Natarajan K, Fong P, Greenspon L, Tamaddon H, Piracha AR, Engelhardt T, Katopodis J, Marques V, Sharp ASP, Piazza G, Goldhaber SZ. A Randomized Trial of the Optimum Duration of Acoustic Pulse Thrombolysis Procedure in Acute Intermediate-Risk Pulmonary Embolism: The OPTALYSE PE Trial. JACC Cardiovasc Interv. 2018 Jul 23;11(14):1401-1410. doi: 10.1016/j.jcin.2018.04.008. PMID 30025734
- [Background] Sharifi M, Bay C, Schwartz F, Skrocki L. Safe-dose thrombolysis plus rivaroxaban for moderate and severe pulmonary embolism: drip, drug, and discharge. Clin Cardiol. 2014 Feb;37(2):78-82. doi: 10.1002/clc.22216. Epub 2013 Oct 7. PMID 24122947
- [Background] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Porcari A, Raskob GE, Weitz JI; AMPLIFY-EXT Investigators. Apixaban for extended treatment of venous thromboembolism. N Engl J Med. 2013 Feb 21;368(8):699-708. doi: 10.1056/NEJMoa1207541. Epub 2012 Dec 8. PMID 23216615
- [Background] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Masiukiewicz U, Pak R, Thompson J, Raskob GE, Weitz JI; AMPLIFY Investigators. Oral apixaban for the treatment of acute venous thromboembolism. N Engl J Med. 2013 Aug 29;369(9):799-808. doi: 10.1056/NEJMoa1302507. Epub 2013 Jul 1. PMID 23808982
- [Background] Rigby RA, Stasinopoulos DM. (2005) Generalized additive models for location, scale and shape. Journal of the Royal Statistical Society: Series C (Applied Statistics). 54(3):507-54.
- [Background] Heo YA. Andexanet Alfa: First Global Approval. Drugs. 2018 Jul;78(10):1049-1055. doi: 10.1007/s40265-018-0940-4. PMID 29926311
- [Background] Vickers AJ. The use of percentage change from baseline as an outcome in a controlled trial is statistically inefficient: a simulation study. BMC Med Res Methodol. 2001;1:6. doi: 10.1186/1471-2288-1-6. Epub 2001 Jun 28. PMID 11459516
- [Background] van Buuren S, Fredriks M. Worm plot: a simple diagnostic device for modelling growth reference curves. Stat Med. 2001 Apr 30;20(8):1259-77. doi: 10.1002/sim.746. PMID 11304741
- [Background] R Core Team (2018). A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated early and never unblinded. Arm/Group randomization information is not available.
Groups:
- All Study Participants: Participants were randomly assigned to either:
  1. Alteplase & Unfractionated Heparin & Apixaban
     Alteplase 24mg intravenous infusion for 20 minutes followed by unfractionated heparin intravenous infusion over 24 hours followed by apixaban 10mg tablet twice-daily for one week followed by apixaban 5mg tablet twice-daily for at least 6 months.
     Alteplase: Lyophilized powder for reconstitution in 50mg vials Unfractionated heparin: Heparin sodium in 0.45% sodium chloride injection for intravenous use Apixaban: Apixaban tablet
     OR
  2. Placebo & Unfractionated Heparin & Apixaban
  Alteplase placebo solution 24mg intravenous infusion for 20 minutes followed by unfractionated heparin intravenous infusion over 24 hours followed by apixaban 10mg tablet twice-daily for one week followed by apixaban 5mg tablet twice-daily for at least 6 months.
  Unfractionated heparin: Heparin sodium in 0.45% sodium chloride injection for intravenous use Placebo: Saline solution reconstituted to mimic Alteplase 50mg vial Apixaban: Apixaban tablet
Period: Overall Study
Arm/Group | All Study Participants
Started | 4
Completed | 3
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The study was closed prematurely due to covid-19. Unblinding was not done and analysis was not performed.
Groups:
- All Study Participants: Participants were randomly assigned to either:
  Alteplase & Unfractionated Heparin & Apixaban Alteplase 24mg intravenous infusion for 20 minutes followed by unfractionated heparin intravenous infusion over 24 hours followed by apixaban 10mg tablet twice-daily for one week followed by apixaban 5mg tablet twice-daily for at least 6 months.
  Alteplase: Lyophilized powder for reconstitution in 50mg vials Unfractionated heparin: Heparin sodium in 0.45% sodium chloride injection for intravenous use Apixaban: Apixaban tablet OR Placebo & Unfractionated Heparin & Apixaban Alteplase placebo solution 24mg intravenous infusion for 20 minutes followed by unfractionated heparin intravenous infusion over 24 hours followed by apixaban 10mg tablet twice-daily for one week followed by apixaban 5mg tablet twice-daily for at least 6 months.
  Unfractionated heparin: Heparin sodium in 0.45% sodium chloride injection for intravenous use Placebo: Saline solution reconstituted to mimic Alteplase 50mg vial Apixaban: Apixaban tablet
Arm/Group | All Study Participants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 62.5 [42 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Extent of Clot Lysis in the Experimental Arm
Description: Change in percentage of clot lysis in the experimental arm only as measured using the Refined Modified Miller Score (RMMS) from the baseline CTA to the 24 hour CTA after 24mg of systemic (IV) tPA + standard anticoagulation therapy (experimental arm).
Time Frame: Baseline, 24 hours
Population: The study was terminated early and never unblinded. Data was not analyzed.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Extent of Clot Lysis Between the Experimental Arm and the Active Comparator Arm
Description: Change in percentage of clot lysis between the experimental arm and the active comparator arm as measured using the Refined Modified Miller Score (RMMS) from the baseline CTA to the 24 hour CTA after 24mg of systemic (IV) tPA + standard anticoagulation therapy (experimental arm) compared to 24mg of systemic (IV) placebo + standard anticoagulation therapy (active comparator arm).
Time Frame: Baseline, 24 hours
Population: Data analysis not done because study closed early due to COVID-19 and there were only 4 subjects enrolled. With only 4 subjects, we decided not to unblind due to the sample size being so small that statistical significance could never be demonstrated.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Right Ventricular to Left Ventricular Diameter (RV/LV) Ratio
Description: RV/LV ratio as measured by chest CTA from baseline to 24 ± 6 hours after the infusion of very low dose systemic (IV) tPA in patients with acute intermediate-high risk PE compared with placebo.
Time Frame: Baseline, 24 hours
Population: as for outcome 2
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in RV/LV Ratio From Baseline Echocardiogram
Description: Change from baseline in echocardiographic parameters as measured by the RV/LV ratio within 24 hours ± 6 hours and at 30 ± 5 days after the end of the systemic (IV) tPA infusion compared with placebo.
Time Frame: Baseline, 24 hours and 30 days
Population: as for outcome 2
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Tricuspid Annular Plane Systolic Excursion (TAPSE) From Baseline Echocardiogram
Description: Change from baseline in echocardiographic parameters as measured by the tricuspid annular plane systolic excursion (TAPSE) within 24 hours ± 6 hours and at 30 ± 5 days after the end of the systemic (IV) tPA infusion compared with placebo.
Time Frame: Baseline, 24 hours and 30 days
Population: as for outcome 2
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Right Ventricular Systolic Pressure (RVSP) From Baseline Echocardiogram
Description: Change from baseline in echocardiographic parameters as measured by the estimated right ventricular systolic pressure (RVSP) within 24 hours ± 6 hours and at 30 ± 5 days after the end of the systemic (IV) tPA infusion compared with placebo.
Time Frame: Baseline, 24 hours and 30 days
Population: as for outcome 2
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in the Collapse of the Inferior Vena Cava (IVC) From Baseline Echocardiogram
Description: Change from baseline in echocardiographic parameters as measured by the collapse of the inferior vena cava (IVC) with respiration within 24 hours ± 6 hours and at 30 ± 5 days after the end of the systemic (IV) tPA infusion compared with placebo.
Time Frame: Baseline, 24 hours and 30 days
Population: as for outcome 2
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in the Requirement for Oxygen Therapy After 6 Minute Walk Test (6MWT)
Description: 6MWT distance as measured by the requirement for oxygen therapy at 30 day, 60 day and one year ± 14 days clinic follow-up compared with placebo.
Time Frame: 30 days, 60 days, and 1 year
Population: as for outcome 2
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Borg Dyspnea Scale Score After 6 Minute Walk Test (6MWT)
Description: 6MWT distance as measured by the Borg Dyspnea Scale score (Borg score) at 30 day, 60 day and one year ± 14 days clinic follow-up compared with placebo. The Borg Scale measures self-reported intensity and severity of breathlessness (dyspnea) and fatigue before, during, and after a 6MWT. Each item is scored 0 - 10 (0 = no breathlessness at all; 10 = most severe breathlessness that you have ever experienced), yielding a total between 0 and 20.
Time Frame: 30 days, 60 days, and 1 year
Population: as for outcome 2
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) Questionnaire
Description: Quality of life (QOL) as measured by the PROMIS PF-6at 30 days, 6 months and one year ± 14 days clinic follow-up compared with placebo. The PROMIS PF-6 measures self-reported physical function for everyday tasks (i.e., yard work, shopping, walking up/down stairs). Each item is score 1 - 5 (1 = unable to do/cannot do; 5 = without any difficulty/not at all), yielding a total between 6 and 30.
Time Frame: 30 days, 6 months, and 1 year
Population: as for outcome 2
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Pulmonary Embolism Quality of Life (PEmb-QOL) Questionnaire
Description: Quality of life (QOL) as measured by the PEmb-QOL at 30 days, 6 months and one year ± 14 days clinic follow-up compared with placebo. The PEmb-QOL measures self-reported QOL after a Pulmonary Embolism. The PEmb-QOL has nine sub-scales with higher scores indicating worse outcomes. Each item is score 1 - 5 (1 = unable to do/cannot do; 5 = without any difficulty/not at all), yielding a total between 6 and 30.
Time Frame: 30 days, 6 months, and 1 year
Population: as for outcome 2
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Recurrent Deep Vein Thrombosis (DVT) and/or Pulmonary Embolism (PE) Events
Description: Measured as the number of recurrent DVT and/or PE events in patients at 30 days, 60 days, 6 months, and 1 year compared to placebo.
Time Frame: 30 days, 60 days, 6 months, and 1 year
Population: as for outcome 2
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 8.5months given patient safety concerns due to the COVID-19 pandemic. The original Adverse Event assessment per the protocol was 1 year from baseline.
Description: Study was not unblinded. All data was entered in the treatment fields.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=4)
AKI and Anemia (Renal and urinary disorders) | 1 (1) — Kidney injury which he also has a long history of since 2015. Found to have anemia with a Hgb of 6.5 (He was given a unit of PRBCs and increased to 8.4). CT abdomen showed no major pathology. He did have fecal impaction at other hospital.
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient experienced respiratory failure and patient's family decided to make him DNR. He was placed in hospice facility and died a few days later.
Anemia (Blood and lymphatic system disorders) | 1 (1) — Found to have anemia with Hgb of 6.5. He was given a unit of PRBC's and increased 8.4.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=4)
Headache (Nervous system disorders) | 1 (1) — Headache after TNK administration
Eye pain (Eye disorders) | 1 (1) — Patient had pain in right eye that was sharp in nature. No loss of vision although patient stated that over the last 6 mo the patient felt slight decreased visual acuity bilaterally.
Stomach pain (Gastrointestinal disorders) | 1 (1)
Suspected bleed (Blood and lymphatic system disorders) | 1 (1) — Unknown drop of hemoglobin requiring transfusion
Bruising on chest (Blood and lymphatic system disorders) | 1 (1)
increased shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Suspected bleed (Blood and lymphatic system disorders) | 1 (1) — seems to be related to ulceration on palate which was noted during hospital stay
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Suspected bleed (Blood and lymphatic system disorders) | 1 (1) — bleeding of gums from toothbrushing
worsening back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — worsening with bending down-- chest CTA showed clot burden in lungs.
left groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) — discomfort in groin that feels like a twisting and jolt
palpitations (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was held and study closed prematurely due to COVID-19 pandemic. We were otherwise hopeful to enroll and complete all assessments for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT03988842/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT03988842/ICF_001.pdf